CLINICAL TRIAL: NCT06932367
Title: The Efficacy of Dexketoprofen And Methylprednisolone in the Acute Low Back Pain
Acronym: Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ali Gur (Other)
Responsible Party: Sponsor-Investigator, Ali Gur, Assoc.Prof., Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.30.2.ATA0.01.00/286; TTU-2021-9373 (Other Grant/Funding Number: Ataturk University)
Record Dates: First submitted 2025-04-07; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
Keywords: Low back pain; Dexketoprofen; Methylprednisolone; Visual Analog Scale; Oswestry Disability Index
MeSH Terms: conditions — Low Back Pain | interventions — dexketoprofen trometamol; Methylprednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Group 1 was the patients who was receiving intravenous dexketoprofen treatment in 100 saline. The efficacy of the treatments received by the patients was evaluated with the VAS at minutes 0, 15, 30, and 60 and hour 48
  Interventions: Drug: Dexketoprofen (KETAVEL 50 mg/2 ml)
- Group 2 (Active Comparator): Group 2 was the patients who was receiving intravenous dexketoprofen combined with methylprednisolone treatment in 100 saline. The efficacy of the treatments received by the patients was evaluated with the VAS at minutes 0, 15, 30, and 60 and hour 48.
  Interventions: Combination Product: Methylprednisolone (Corticosteroid)

INTERVENTIONS:
Drug: Dexketoprofen (KETAVEL 50 mg/2 ml) — Patients with low back pain were divided in to two groups: those receiving intravenous dexketoprofen treatment (Group 1) and those receiving dexketoprofen + methylprednisolone treatment (Group 2). The efficacy of the treatments received by the patients was evaluated with the VAS at minutes 0, 15, 30, and 60 and hour 48. Statistical evaluations were also undertaken on the ODI results evaluated at minute 0 and hour 48.
  Arms: Group 1
Combination Product: Methylprednisolone (Corticosteroid) — Patients with low back pain were divided in to two groups: those receiving intravenous dexketoprofen treatment (Group 1) and those receiving dexketoprofen + methylprednisolone treatment (Group 2). The efficacy of the treatments received by the patients was evaluated with the VAS at minutes 0, 15, 30, and 60 and hour 48. Statistical evaluations were also undertaken on the ODI results evaluated at minute 0 and hour 48.
  Arms: Group 2

SUMMARY:
Many methods have been used in to treat low back pain. In this study, we aimed to investigate the efficacy of dexketoprofen alone and in combination with methylprednisolone in the treatment of low back pain in the emergency department using the Visual Analog Scale (VAS) and the Oswestry Disability Index (ODI).This prospective, randomized, single-blind study included 150 patients admitted to the emergency department of a university hospital. Patients with low back pain were divided in to two groups: those receiving intravenous dexketoprofen treatment (Group D) and those receiving dexketoprofen + methylprednisolone treatment (Group DM). The efficacy of the treatments received by the patients was evaluated with the VAS at minutes 0, 15, 30, and 60 and hour 48. Statistical evaluations were also undertaken on the ODI results evaluated at minute 0 and hour 48.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 and under 65 years.
* The patients who presented to the emergency department with acute non-traumatic low back pain.
* Voluntarily agreed to participate in the study.

Exclusion Criteria:

* The patients who had used analgesics within the last six hours;
* Who has neurological deficits, cardiac or chest pain, liver, kidney, cardiac or pulmonary failure, chronic pain,
* Who has a history of dexketoprofen-related gastrointestinal bleeding or perforation, referred pain, neoplastic pain, a history of allergies to medications used in the study (methylprednisolone and dexketoprofen), or vision problems;
* Who indicated a pain intensity of 3 cm or less on the 10-cm VAS scale line at the time of their presentation to the emergency department; pregnant and breastfeeding women;
* The patients who were illiterate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) score | 48 hours
  The primary outcome of the study was the pain scores of the groups according to the Visual Analog Scale (VAS) scores. Lower VAs score below 4 is assigned as the lower pain value of the participants, whereas, higer vaslus of VAS score close to 10 accepted as higher pain value described from the participants

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 48 hours
  The secondary outcome was the effect of dexketoprofen alone and in combination with methylprednisolone on low back pain-related disability, according to the Oswestry Disability Index (ODI)scores.
  While interpreting the ODI score, the the scores are considered as:
  0% to 20% - minimal disability 20% to 40% - moderate disability 40% to 60% - severe disability 60% to 80% - crippled 80% to 100% - bed bound (or exaggerating symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Meral Ataturk University Medical Faculty, Emergency Department, M.D., Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author, upon reasonable request.

REFERENCES:
- [Derived] Meral M, Gur A. A comparative study on the efficacy of dexketoprofen and methylprednisolone in the treatment of acute low back pain. BMC Emerg Med. 2025 Aug 5;25(1):147. doi: 10.1186/s12873-025-01276-y. PMID 40765043